CLINICAL TRIAL: NCT02237339
Title: Does Allopurinol Regress Left Ventricular Hypertrophy in Patients With Treated Essential Hypertension?
Brief Title: Does Allopurinol Reduce Thickening of the Left Ventricle of the Heart in Patient With Treated Hypertension?
Acronym: ALLAY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012CV15; 2014-002083-33 (EudraCT Number)
Record Dates: First submitted 2014-08-18; First posted 2014-09-11 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Hypertension; Hypertrophy, Left Ventricular
Keywords: Allopurinol; Cardiac MRI (CMR); Flow mediated dilatation (FMD); Pulse wave analysis (PWA); Endothelial function; Scar; Hypertrophy; Hypertension
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular; Cicatrix; Hypertrophy | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol (Active Comparator): Patients treated with Allopurinol 300mg daily for first month then 300mg twice daily for remainder trial.
  Interventions: Drug: Allopurinol
- Placebo tablet (Placebo Comparator): Microcrystalline cellulose one tablet daily for first month then twice daily for remainder of trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — Uric acid lowering medication.
  Other Names: Zyloric
  Arms: Allopurinol
Drug: Placebo
  Arms: Placebo tablet

SUMMARY:
The presence of Left ventricular hypertrophy (LVH) confers high cardiovascular risk in hypertensive patients. LVH remains highly prevalent even when blood pressure (BP) is controlled. There is increasing evidence that a major non-haemodynamic contributor to LVH is oxidative stress. Allopurinol is known to markedly reduce oxidative stress.

This pragmatic randomised double blind placebo controlled trial will examine whether allopurinol (300 mg bd) regresses LV mass as assessed by cardiac magnetic resonance (CMR) in 66 patients with treated hypertension but who have persisting LVH.

Endothelial and vascular function will also be assessed via flow mediated dilatation (FMD) and pulse wave analysis respectively (PWA) and plasma biomarkers of oxidative stress will be measured. The treatment (allopurinol or placebo) will last 12 months.

DETAILED DESCRIPTION:
Does Allopurinol regress Left Ventricular Hypertrophy in Patients with Treated Essential Hypertension?

People with high blood pressure are at increased risk of heart complications. One of the biggest problems is that the muscle wall of the heart thickens. The medical term for this is Left Ventricular Hypertrophy (LVH). LVH makes the heart less efficient and patients with LVH are at a 10 times greater risk of heart complications than those without it.

A goal of treating high blood pressure is to reduce the strain on the heart and to try to decrease this thickening of the heart wall. However, even when blood pressure is treated and is under control, LVH can persist, and as there are no symptoms to LVH it can go undetected.

Currently the only way to reduce LVH would be to lower blood pressure (BP) even further. This can cause side-effects from low BP such as dizziness and nausea.

It has previously been shown that a drug allopurinol, which is usually used to treat gout had the remarkable side effect of being able to reduce this thickening of the heart wall in patients who had kidney disease or diabetes. The aim now is to see if patients with high blood pressure and LVH may also benefit from treatment with allopurinol. If LVH can be reduced using allopurinol, this might be a new way to reduce cardiac risk in these patients without needing to lower BP even further.

In this study the aim is to recruit 66 patients who have treated and well controlled blood pressure but may still have LVH. They will be screened for LVH by doing an ultrasound scan of the heart and then that will be confirmed with a Magnetic Resonance Imaging (MRI) scan, which is a special scan of the heart using an MRI machine to measure the extent of thickening of the heart muscle before they start on treatment of allopurinol or placebo.

As this is a clinical trial the participants will be randomly allocated to either allopurinol or a dummy medication (placebo) and will receive one year of treatment so that the investigators can compare if there is a difference between normal treatment and addition of allopurinol. All the patients currently prescribed medication for their high blood pressure will continue as normal on that. They will have a further MRI scan when their one year treatment with allopurinol or placebo finishes.

Benefits - You will be monitored closely during the study and will be seen by a doctor with a special interest in cardiology at each of your study visits and your medication will be reviewed on a regular basis. The tests will give us information about the function of your heart, kidneys and blood circulation. If any of these investigations, including information from the MRI scan of your heart reveal any new abnormality we will either discuss this with your hospital consultant or refer you to a specialist clinic (whichever seems most appropriate). The study will not immediately benefit you, but if the results of the study are positive it may change the practice of managing patients with treated high blood pressure but may still have LVH, like you and potentially will have a great impact on other such patients in the future. If so, you may gain eventually from our discovering a new treatment for your condition.

Risks - The side effects of the allopurinol are very rare (less than 1 in 10,000 people) and include headache, stomach upset, drowsiness and anaemia. Having blood tests taken can cause some mild bruising. The flow mediated dilatation may cause temporary numbness. MRI scanning is very safe and does not use radiation but some may feel a bit closed in. The scanner is a bit noisy but you will be given ear protection which also plays music. Your kidney function will be assessed before the scan to ensure it is safe to give you the contrast agent described above.

ELIGIBILITY:
Inclusion Criteria:

* are aged over 18 years
* previously diagnosed with essential hypertension
* been on stable antihypertensive therapy for at least 3 months prior to study screening
* have screening ambulatory bloods pressure monitoring (ABPM) or home based BP monitoring if ABPM not tolerated with daytime average systolic <135mmHg
* have screening echocardiography based diagnosis of left ventricular hypertrophy (LVH) based on American society of echocardiography (ASE) criteria (males >115g/m2, females >95g/m2)

Exclusion Criteria:

* documented intolerance to allopurinol
* left Ventricular Ejection Fraction <45% on echocardiography screening
* severe aortic stenosis on echocardiography screening
* active gout (i.e. flare within two years) or currently on allopurinol
* severe hepatic disease
* renal disease; chronic kidney disease (CKD) class 3B or worse
* on azathioprine, 6 mercaptopurine, or theophylline
* malignancy (receiving active treatment) or other life threatening diseases
* pregnant or lactating women
* any contraindication to magnetic resonance imaging (MRI) (claustrophobia, metal implants, penetrative eye injury or exposure to metal fragments in eye requiring medical attention).
* patients who have participated in any other clinical trial of an investigational medicinal product within the previous 30 days will be excluded.
* patients who are unable to give informed consent
* any other considered by a study physician to be inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The change LV mass index with allopurinol versus placebo. | 12 months
  Baseline and repeat CMRI examinations at baseline (+/- 2 weeks) and after the final 12 month (+/- 2 weeks) visit will be performed on a 3T Magnetom scanners (Siemens, Erlangen, Germany) using dedicated phase array cardiac coils.
  Analysis will be performed offline (Argus Software, Siemens) by a single blinded observer for the assessment of left ventricular mass. This single observer will analyze all the scans. The reproducibility of the left ventricular mass assessment using MRI will be derived for this observer.
  The change LV mass index in participants treated with allopurinol will be compared with placebo.

SECONDARY OUTCOMES:
% change in brachial artery diameter and change in augmentation index with allopurinol versus placebo. | 12 months
  Flow mediated dilatation (FMD) of the brachial artery will be performed on two visits (baseline and month 12) according to the guide-lines set by the International Brachial Artery Reactivity Task Force. FMD will be expressed as percent change in diameter relative to the baseline diameter at rest. Analysis of all FMDs will be performed on Brachial Analyser software by a single trained investigator. This investigator will be blind to allocated treatments.
  . PWA and PWV will be determined in the arm by recording the radial waveforms and radial-carotid waveforms, respectively, at two visits (baseline and month 12) using the Sphygmocor system. The central augmentation index (AIx) will be corrected to a heart rate of 75 beats/min. A single trained investigator who is blind to the allocated treatment will perform the PWA and PWV.
Change in average 24 hour BP control with allopurinol versus placebo. | 12 months
  Patient will undergo 24 hour ambulatory BP monitoring after the screening and final visit (12 months) to assess the difference in blood pressure control with allopurinol versus placebo.
The change in C reactive protein (CRP), brain natriuretic peptide (BNP), troponin I (TnI), oxidized lactate dehydrogenase (oxidized LDH) and Procollagen carboxyl end peptide (PICP) with allopurinol versus placebo. | 12 months
  Research bloods will be taken at vist 2 (day 0) and visit 7 (12months) and will compare changes between groups.
Measure a change in left ventricular (LV) mass, LV end systolic volume, LV end diastolic volume or LV ejection fraction. | Twelve months
  Baseline and repeat CMRI examinations at baseline (+/- 2 weeks) and after the final 12 month (+/- 2 weeks) visit will be performed on a 3T Magnetom scanners (Siemens, Erlangen, Germany) using dedicated phase array cardiac coils.
  Analysis will be performed offline (Argus Software, Siemens) by a single blinded observer for the assessment of ventricular volumes (EDV, ESV, stroke volume), EF, and left ventricular mass. This single observer will analyze all the scans.
  The reproducibility of the left ventricular mass assessment using MRI will be derived for this observer.
  We will assess left ventricular (LV) mass, LV end systolic volume, LV end diastolic volume and LV ejection fraction in participants treated with allopurinol versus placebo.
The change in LV mass after subtracting the volume of scar with allopurinol versus placebo. | 12 months
  Baseline and repeat CMRI examinations at baseline (+/- 2 weeks) and after the final 12 month (+/- 2 weeks) visit will be performed on a 3T Magnetom scanners (Siemens, Erlangen, Germany) using dedicated phase array cardiac coils.
  Analysis will be performed offline (Argus Software, Siemens) by a single blinded observer for the assessment of left ventricular mass and scar volume.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gingles, MBChB, Principal Investigator — University of Dundee; Jacob George, MBChB, Study Director — University of Dundee
Locations (1):
- University of Dundee, Ninewells Hospital, Dundee, Tayside, United Kingdom

REFERENCES:
- [Derived] Gingles CR, Symon R, Gandy SJ, Struthers AD, Houston G, MacDonald TM, Lang CC, Donnan PT, George J. Allopurinol treatment adversely impacts left ventricular mass regression in patients with well-controlled hypertension. J Hypertens. 2019 Dec;37(12):2481-2489. doi: 10.1097/HJH.0000000000002189. PMID 31268872